CLINICAL TRIAL: NCT06737081
Title: A Parallel, Open-label Phase II Clinical Study of Enarodustat (SAL-0951) Tablets in the Treatment of Chemotherapy-induced Anemia in Patients With Non-myeloid Malignancies
Brief Title: SAL-0951 in the Treatment of Chemotherapy-induced Anemia in Patients With Non-myeloid Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAL0951B201
Record Dates: First submitted 2024-12-04; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Anemia
Keywords: Chemotherapy; Anemia; Enarodustat
MeSH Terms: conditions — Anemia | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAL-0951 tablets 4mg (Experimental): initial phase：4mg QD subsequent phase：1mg～8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: SAL-0951 tablets 4mg
- SAL-0951 tablets 5mg (Experimental): initial phase：5mg QD subsequent phase：1mg～8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: SAL-0951 tablets 5mg

INTERVENTIONS:
Drug: SAL-0951 tablets 4mg — initial phase：4mg QD subsequent phase：1mg～8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Other Names: SAL-0951 tablets 4mg group
  Arms: SAL-0951 tablets 4mg
Drug: SAL-0951 tablets 5mg — initial phase：5mg QD subsequent phase：1mg～8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Other Names: SAL-0951 tablets 5mg group
  Arms: SAL-0951 tablets 5mg

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of SAL-0951 in the treatment of chemotherapy-induced anemia (CIA) in patients with non-myeloid malignancies

DETAILED DESCRIPTION:
This trial is a multicenter, randomized, open-label phase II clinical study exploring the starting dose, aiming to evaluate the safety and efficacy of Enarodustat Tablets in the treatment of chemotherapy-induced anemia (CIA) in patients with non-myeloid malignancies, so as to optimize the dose for phase III trials. It is planned to enroll approximately 60 patients.

The trial consists of a screening period (4 weeks), an open-label treatment period (up to 16 weeks), and a follow-up period (2 weeks), totaling approximately 22 weeks. Subjects who withdraw early will be asked to complete an end of treatment visit, and a safety follow-up visit 2 weeks after the end of treatment visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with body weight ≥40 kg at screening;
2. Subjects with histologically or cytologically confirmed diagnosis of non-myeloid malignancy (non-curative), and planned to receive anti-tumor treatment (myelosuppressive chemotherapy) for at least 6 weeks simultaneously from the day of the first dose (Day 1);
3. Subjects with myelosuppressive chemotherapy-related anemia, defined as central laboratory Hb ≤100 g/L during the screening period, and documented decrease in Hb level ≥10 g/L after the start of chemotherapy as judged by the investigator;
4. Subjects with ferritin ≥50 ng/mL and transferrin saturation (TSAT) ≥10% at screening;
5. Subjects with Eastern Cooperative Oncology Group (ECOG) performance status score ≤1 at screening;
6. Subjects with life expectancy ≥6 months as judged by the investigator on the date of first dose;
7. All male subjects and female subjects of childbearing potential who agree to use a medically acceptable method of contraception from the day of signing the ICF until 90 days after last dose of investigational product (see section 4.3 for acceptable method of contraception);
8. Subjects voluntary to participate in the trial, having signed the ICF, able to understand the procedures and methods of this trial and willing to strictly follow the clinical trial protocol to complete the trial.

Exclusion Criteria:

1. Subjects with tumor who are receiving myelosuppressive chemotherapy and whose expected outcome is cured;
2. Subjects who receive hormonal agents, biologics, novel immunosuppressants (e.g., PD-1 and PD-L1 immune checkpoint inhibitors) or targeted biologic therapy or radiation therapy alone to treat/control their tumors. However, if chemotherapy is used in combination with these drugs, subjects can be enrolled;
3. Subjects who have received blood transfusion therapy containing red blood cells or ESAs (including but not limited to recombinant human erythropoietin, darbepoetin alfa, methoxy polyethylene glycol-epoetin beta/CERA, pegmolesatide) within 4 weeks before the first dose of investigational product;
4. Subjects with abnormal hepatic or renal function test results at screening as follows:

   * Patients with alanine transaminase (ALT) >3×upper limit of normal (ULN), or aspartate transaminase (AST) >3×ULN, or total bilirubin (TBL) >1.5×ULN are not allowed to be enrolled in the study (those with TBL ≤2×ULN can be included if ALT/AST is within the normal limit and the investigator believes that there is no safety concern)
   * With estimated glomerular filtration rate (eGFR) of <30 mL/min/1.73 m2 based on CKD-EPI 2009scr formula, as shown in Appendix 3.
5. Subjects with congestive heart failure (New York Heart Association [NYHA] Class III or greater), unstable angina, uncontrolled hypertension (defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg despite antihypertensive medication), or hypertensive crisis or hypertensive encephalopathy, or a history of significant valvular or endocardial disease that would put them at risk for thromboembolism within 6 months prior to screening and/or within the screening period;
6. Subjects with thromboembolic events (including but not limited to deep vein thrombosis [DVT], pulmonary embolism, myocardial infarction, stroke, transient ischemic attack [TIA]) within 6 months prior to screening (excluding asymptomatic lacunar infarction);
7. Subjects with clinically significant anemia caused by other causes, such as macrocytic anemia caused by vitamin B12 or folic acid deficiency, autoimmune anemia, hemolysis, genetic anemia such as sickle cell anemia or thalassemia, anemia caused by severe infection (such as active pulmonary tuberculosis, fungal infection, etc.) or existing active bleeding lesions (such as lung cancer-related hemoptysis, gastrointestinal tumor bleeding, gastrointestinal ulcer bleeding, etc.);
8. Subjects with active systemic infection requiring chronic antibiotic therapy;
9. Subjects with clinically significant or uncontrolled ongoing inflammatory/autoimmune disease (e.g., systemic lupus erythematosus, rheumatoid arthritis, Crohn's disease, celiac disease, etc.);
10. Subjects with need for an ophthalmological procedure due to diabetic eye disease, diabetic macular edema or age-related macular degeneration, or subjects with proliferative choroidal or retinal lesions;
11. Subjects known to have significant gastrointestinal abnormalities, which would affect drug intake, transport or absorption (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or total gastrectomy;
12. Subjects known to have polycystic kidney disease;
13. Subjects known to have serious liver disease or active liver disease (except non-alcoholic hepatic steatosis), including chronic hepatitis B (positive for hepatitis B surface antigen or hepatitis B core antibody, and HBV-DNA >20 IU/mL), chronic hepatitis C (positive for hepatitis C antibody, and HCV-RNA quantitative detection higher than the upper limit of normal), autoimmune hepatitis, cirrhosis, or acute liver failure;
14. Subjects tested positive for human immunodeficiency virus (HIV) antibody;
15. Subjects with major surgery anticipated to occur during the trial;
16. Subjects with myeloid malignancies (such as chronic myeloid leukemia, etc.);
17. Subjects with primary or metastatic malignant tumors of the central nervous system;
18. Subjects with anticipated use of dapsone during the trial;
19. Subjects with hypersensitivity to HIF-PH inhibitors or any of the product components;
20. Subjects with a history of drug or alcohol abuse in the past two years*;

    *An average of 14 units of alcohol per week (1 unit ≈ 360 mL of beer, or 45 mL of liquor, or 150 mL of wine) in 2 years before screening.
21. Subjects who have received another investigational product (or study drug), have received treatment with an investigational device (or study device), or have participated in clinical research involving intervention (medical action beyond the scope of ordinary medical practice) and received treatment during the period within 8 weeks prior to the screening;
22. Subjects who have participated in clinical trials of HIF-PH inhibitor treatment (including enarodustat) within 4 weeks before screening and have received investigational product (active drug) treatment;
23. Subjects who are pregnant, lactating, or may be pregnant (the possibility of pregnancy cannot be ruled out by the investigator based on the results of pregnancy test at screening visit);
24. Subjects who have taken traditional Chinese medicine, Chinese patent medicine, and/or herbal medicine for anemia within 2 weeks before the first dose of investigational product;
25. Subjects with any other medical condition that, in the opinion of the investigator, could pose a safety risk to them in this trial, could confound efficacy or safety assessment, or could interfere with their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events by CTCAE5.0 | through study completion, an average of 4 months
  laboratory abnormalities (based on whole blood count, biochemistry, coagulation function, fecal occult blood test and urinalysis tests), vital sign measurements (include blood pressure, pulse rate and body-temperature), physical examination-and-12-Lead electrocardiogram.

SECONDARY OUTCOMES:
Change from baseline in mean Hb at the end of treatment (EOT); | through study completion, an average of 4 months
  through study completion, an average of 4 months, the change from baseline in mean Hb at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No